CLINICAL TRIAL: NCT02820376
Title: Assessment of Differential Renal Function by CT in Living Donors - The DOVISCAN Study
Brief Title: Assessment of Differential Renal Function by CT in Living Donors
Acronym: DOVISCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A00543-48; PSS 2016 / DOVISCAN - MANDRY / (Other: CentralHNF)
Record Dates: First submitted 2016-06-20; First posted 2016-07-01 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Living Donor of Kidney
Keywords: 4D computed tomography; Kidney function tests; Living Donors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Other): Differential renal function assessment by 4D CT:
  All patients will undergo both CT and SPECT assessment of differential renal function; each patient will be his own comparator
  Interventions: Other: Differential renal function assessment by 4D CT

INTERVENTIONS:
Other: Differential renal function assessment by 4D CT — Low dose 4D (perfusion) renal acquisition after injection of iodinated contrast medium (ICM) (13 passes every 3 seconds, 3 passes every 10 seconds); estimated additional DLP 400 mGy.cm No additional contrast medium

SUMMARY:
The purpose of this study is to assess the degree of agreement of the measurement of differential renal function in living donors by CT (computed tomography) and SPECT (single photon emission computed tomography).

ELIGIBILITY:
Inclusion Criteria:

* Kidney living donor candidate (approval given) undergoing a morphological and functional renal assessment
* Mandatory enrollment in a health security plan (French Social Security)
* Subject having signed an informed consent

Exclusion Criteria:

* Contra-indications to computed tomography with iodinated contrast medium injection, or to scintigraphy
* Subjects with an abnormal urinary tract (unique kidney, ectopic kidney, horseshoe kidney)
* Subjets under a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
degree of agreement | through study completion (2 years)
  Differential renal function (DRF) measured by each technique (CT and SPECT) Regions of interest will be drawn on each kidney and the aorta to obtain time-intensity curves and derive the Patlak plot; the Patlak model will then be used to determine the slope of each kidney and thus to calculate the differential renal function (percentage of each kidney in the total renal function).
  Degree of agreement will be assessed by calculating the intra-class correlation coefficient and its 95% confidence interval, and the Bland-Altman plot.

SECONDARY OUTCOMES:
Intra- and inter-observer reproducibility of CT DRF measurement | through study completion (2 years)
Radiation dose exposure for each technique | 1 day
  Additional radiation dose exposure (CTDIvol and DLP) will be recorded and follow-up
Agreement between post-processing methods for CT | through study completion (2 years)
  Comparison between Patlak-Ruthland method, its modified version and the area under the curve method
Automatic post-processing for Patlak-Ruthland method | through study completion (2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Damien Mandry, MD,PhD, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No